CLINICAL TRIAL: NCT02998801
Title: Alleviating Pre-operative Anxiety With Innovative 3D Immersive Virtual Reality
Acronym: VR-Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 484-2015
Record Dates: First submitted 2016-11-21; First posted 2016-12-20 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Virtual Reality; Anxiety; Preoperative Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Watch video using IPAD (Placebo Comparator): Patient will watch the educational video using an IPAD
  Interventions: Other: IPAD
- Watch video using VR goggles (Active Comparator): Patient will watch the educational video using VR goggles
  Interventions: Other: VR Goggles

INTERVENTIONS:
Other: IPAD — Patients undergoing surgery will watch the video using an PAD
  Arms: Watch video using IPAD
Other: VR Goggles — Patients undergoing surgery will watch the video using goggles
  Arms: Watch video using VR goggles

SUMMARY:
To construct and evaluate an immersive 3D simulation to familiarize patients with the pre-operative experience, and investigate whether A) immersive 3D virtual reality video can reduce pre-operative anxiety, and B) how this approach compares to current practice of viewing traditional educational videos.

DETAILED DESCRIPTION:
The prevalence of pre-operative anxiety is estimated as being as high as 80% in surgical populations. Physiologically, this may result in higher cortisol levels, which may slow down the healing and recovery process. A multitude of perioperative clinical trials have revealed that pre-operative anxiety is associated with reduced short-term postoperative recovery, increased pain scores, nause & vomiting, sleep disturbances, surgical wound infections, increased length of stay, and cardiac complications. It has also been linked with worse functional outcomes and quality of life up to one-year after surgery.

Literature looking at factors associated with preoperative anxiety outline a general theme of the fear of the unknown that is distressing. Specifically, the most distressing events seem to be waiting to be collected for surgery, waiting outside the operating room (OR), being transferred to the OR bed and having monitors and oxygen mask applied. These moments prior to surgery are when patients are most likely to continuously ruminate over 'what comes next' and the fact of not knowing - leading to anxiety. One survey of 161 patients presenting for elective surgery inquired about factors that led to being calm prior to their procedure and found that being well informed of the pre-operative process was a critical aspect of anxiety relief. Approaches such as implementation of the pre-anesthetic clinic (PAC) and the use of videos of what to expect leading up to surgery have been implemented to address this issue but have been costly or have had mixed effects.

Virtual reality (VR) technology presents a new educational opportunity for patients in an effort to reduce pre-operative anxiety. Through immersive 3D simulation, patients can experience the journey of being prepped for surgery and transferred to the OR. A patient can learn about their pre-operative experience in a more engaging manner as opposed to passively reading, watching video or being verbally taught about it by the healthcare provider. A patient is educated by having the perception of being physically present in the pre-operative experience days or weeks prior to their OR date.

ELIGIBILITY:
Inclusion Criteria:

* All participants less than 80 years old presenting to the pre-assessment clinic at Sunnybrook Health Sciences Centre
* Planned surgical procedure is 7-14 days after pre-assessment clinic visit

Exclusion Criteria:

* Inability to provide informed consent
* Unable to complete study assessments (ie: visually impaired)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Change in anxiety levels as measured using VAS score from baseline to the day of surgery inside the OR. | 2 weeks

SECONDARY OUTCOMES:
Change in heart rate between patients randomized to IPAD or VR Goggles from baseline to the day of surgery inside the OR. | 2 weeks
Change in blood pressure between patients randomized to IPAD or VR Goggles from baseline to the day of surgery inside the OR. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Alam, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided